CLINICAL TRIAL: NCT05874856
Title: Heart Rate Variability, Physical Activity and Exhaustion in the Inpatient Treatment of Stress-Related Disorders
Acronym: HARMODI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Arno Schmidt-Trucksäss (Other)
Responsible Party: Sponsor-Investigator, Arno Schmidt-Trucksäss, Prof. Dr. med. Arno Schmidt-Trucksäss, University of Basel
Organization: University of Basel (Other)
Other Study IDs: 2022-01871
Record Dates: First submitted 2023-02-08; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Depression; Burnout; Stress Related Disorder
Keywords: Stress Related Disorder; Heart Rate Variability; Physical Activity; Exhaustion; Inpatient Treatment; Cardiorespiratory fitness
MeSH Terms: conditions — Depression; Burnout, Psychological; Motor Activity | interventions — Blood Pressure; Pulse Wave Analysis; Cardiorespiratory Fitness; Sleep

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Heart rate variability, blood pressure and pulse wave velocity — Resting HRV in supine and standing position, blood pressure and pulse wave velocity in supine position at first and last week of inpatient treatment
Diagnostic Test: Assessment of cognitive function, balance, strength and cardiorespiratory fitness — THINC-it test for cognitive function; One-leg Standing test for balance assessment; 10-time chair rise test and hand grip test for strength assessment; Åstrand-Ryhming Test for cardiorespiratory fitness.
  All assessments will be performed at first and last week of inpatient treatment.
Behavioral: Monitoring of physical activity and sleep — GENEActiv accelerometer will be worn on the wrist daily during 8-week inpatient treatment.
Behavioral: Monitoring of self-rated exhaustion, mood and tension — Using the customized PsyMate app.

SUMMARY:
The goal of this observational study is to learn about heart rate variability and physical activity in inpatients with stress-related disorder. The main questions to answer are:

* whether heart rate variability shows the severity of certain symptoms.
* whether physical activity has an influence on heart rate variability and symptoms of stress-related disorder.

Participants will be asked to take part in 5 examinations during their up to 8-week inpatient treatment:

* Participate in an interview
* Measurement of heart rate variability, blood pressure and health of the arteries (pulse wave velocity)
* Tests of endurance, strength, balance and cognitive abilities
* Completion of two additional short questionnaires
* Wearing a 24-hour electrocardiogram
* Wearing a fitness watch and daily self-assessment of fatigue, mood and tension via an app on participant's mobile phone during their stay.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of an ICD-10 depressive episode (F32 or F33) and burnout (Z73) without psychotic symptoms
* German language skills
* mobile phone ownership
* age 18-35 years

Exclusion Criteria according to medical history:

* comorbid psychiatric disorder, including post-traumatic stress disorder as well as anxiety and panic disorder
* current treatment with antiarrhythmic drugs and tricyclic antidepressant medication
* factors precluding submaximal endurance test: history of cardiac diseases such as myocardial infarction, stroke and unstable heart failure within the previous six months impairing exercise testing and training, and heart failure (New York Heart Association functional class III and IV)
* factors severely affecting HRV parameters: type 1 & 2 diabetes mellitus with clinically proven cardiovascular autonomic neuropathy, chronic obstructive pulmonary disease Global Initiative for Obstructive Lung Disease stage ≥ III, ongoing cancer treatment, moderate to severe chronic kidney disease (estimated Glomerular Filtration Rate stage 3a (G3a) or worse (≤ 45 ml/min)), current eating disorders such as anorexia nervosa and bulimia nervosa, excessive drug or alcohol abuse
* known pregnancy
* suicidal thoughts precluding informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited among patients referred to the rehabilitation clinic with the diagnosis of an ICD-10 depressive episode (F32 or F33) and burnout (Z73), confirmed by experienced psychiatrists working in the clinic.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Orthostatic Test Heart Rate Variability (HRV) at 8 weeks. | Orthostatic Test HRV will be measured in the first and last week of up to 8-week inpatient treatment.
  Particular focus is RMSSD in milliseconds, a robust parasympathetic nervous system parameter that is less influenced by body movement and breathing.
Change from Baseline 24-hour Heart Rate Variability (HRV) at 8 weeks. | 24-hour HRV will be measured in the first and last week of up to 8-week inpatient treatment.
  Particular focus is RMSSD in milliseconds, a robust parasympathetic nervous system parameter that is less influenced by body movement and breathing.
Change from Baseline Exercise Test Heart Rate Variability (HRV) at 8 weeks. | Exercise Test HRV will be measured in the first and last week of up to 8-week inpatient treatment.
  Particular focus is RMSSD in milliseconds, a robust parasympathetic nervous system parameter that is less influenced by body movement and breathing.

SECONDARY OUTCOMES:
Change from baseline cardiorespiratory fitness at 8 weeks. | Cardiorespiratory fitness will be measured in the first and last week of up to 8-week inpatient treatment.
  Calculated maximal oxygen uptake (VO2max) in (ml/kg/min) based on submaximal testing (Åstrand-Ryhming Test).
Global score of the Hamburger Burnout Inventory (HBI) to assess the severity of the burnout syndrome. | Severity of Burnout syndrome will be measured in the first week of up to 8-week inpatient treatment.
  One item of the 40-item Hamburger Burnout Inventory (HBI) represents a global score on the severity of crisis, which can be rated on a 9-point Likert scale. The Global score can range between 1 and 9, with higher scores indicating worse outcome (worse severity): 1-3 harmless, 4-6 medium and 7-9 need for action.
Total score of the Shirom-Melamed-Burnout-Measure (SMBM) will be used measure exhaustion at the beginning of inpatient treatment. | Exhaustion will be measured in the first week of up to 8-week inpatient treatment.
  Exhaustion with the three dimensions physical, emotional and cognitive exhaustion will be self-rated on a 7-point Likert scale, ranging from 1 (never) to 7 (always). A total score can vary between 14 and 98, with higher scores reflecting a higher degree of exhaustion / worse outcome.
Depression severity will be evaluated with a total score of the German version of the 21-item Beck Depression Inventory-II. | Depression severity will be measured in the first and last week of up to 8-week inpatient treatment.
  Participants will rate their depressive symptoms over the past two weeks on a 4-point Likert scale. Cut-off scores for patients diagnosed with an affective disorder are calculated by the sum of the total score: 0-10 indicates minimal depression, 10-18 mild to moderate depression, 19-29 moderate to severe depression and 30-63 severe depression.
Change of Vital exhaustion with a total score of the 9-item short form of the original 21-item Maastricht Vital Exhaustion Questionnaire (MVEQ). | Vital exhaustion will be measured in the first and last week of up to 8-week inpatient treatment.
  Participants will report whether they feel exhausted 0 (no), 1 (uncertain) and 2 (yes), with a total score ranging from 0 to 18; with 4-10 indicating mild, 11-14 substantial and 15-18 severe vital exhaustion.
Anxiety severity will be displayed with a total score of the 21-item Beck Anxiety Inventory. | Anxiety severity will be measured in the first and last week of up to 8-week inpatient treatment.
  The 21-item Beck Anxiety Inventory (BAI) will assess anxiety symptoms of the last seven days on a 4-point Likert scale ranging from 0 (not at all) to 3 (severely). A total score can vary between 0 to 63, with 0-7 points indicating minimal anxiety, 8-15 mild, 16-25 moderate and 26-63 clinical anxiety.
Mood with a total score of the 14-item German version of the Snaith-Hamilton-Pleasure Scale. | Mood will be measured in the first and last week of up to 8-week inpatient treatment.
  The Snaith-Hamilton-Pleasure Scale (SHAPS-D) will be used to assess self-reported mood on a 4-point Likert scale ranging from "I fully agree" to "I do not agree at all". The participants are asked, related to the last days, to imagine if they feel pleasure in different situations, with a higher total score, ranging between 0 and 14, indicating increased anhedonia.
Current mood will be shown in total scores of the Multidimensional Mood Questionnaire. | Current mood will be measured in the first and last week of up to 8-week inpatient treatment before the HRV measurement.
  The Multidimensional Mood Questionnaire is a self-rated questionnaire (5-Point Likert Scale) with three dimensions: good-bad mood, alertness-fatigue and calmness-restlessness, with high scores (range between 4 and 20) indicating a positive direction, good mood, alertness and calm state.
Daily tiredness displayed with a daily score rated with the single item "How tired do you feel at the moment?" | Level of tiredness daily during up to 8-week inpatient treatment
  The item "How tired do you feel at the moment?" is an adapted version of one item of the Multidimensional Mood Questionnaire. Participants rate on a 5-Point Likert scale ranging from 1 (not at all) to 5 (completely) how physical tired they feel at the end of the day to capture symptom fluctuations throughout inpatient treatment, with higher scores indicating worse outcome (worse tiredness).
Daily mentally exhaustion displayed with the score rated with the single item "How mentally exhausted do you feel at the moment?". | Level of mentally exhaustion daily during up to 8-week inpatient treatment
  The item "How mentally exhausted do you feel at the moment?" is adapted from the German version of the Perceived Stress Questionnaire.
  Participants rate their answers on a 5-point Likert scale ranging from 1 (not at all) to 5 (completely) to capture symptom fluctuations throughout inpatient treatment, with higher scores indicating worse outcome (worse mentally exhaustion).
Daily tension level will be measured with a daily score rated with the single item "How tense do you feel at the moment?". | Level of tension daily during up to 8-week inpatient treatment
  The item "How tense do you feel at the moment?" is adapted from the German version of the Perceived Stress Questionnaire. Participants rate their answers on a 5-point Likert scale ranging from 1 (not at all) to 5 (completely) to capture symptom fluctuations throughout inpatient treatment, with higher scores indicating worse outcome (higher tension).
Total score of the self-rated 5-item Perceived Deficits Questionnaire. | Cognitive function will be self-rated in the first and last week of up to 8-week inpatient treatment.
  The abbreviated 5-item version of the Perceived Deficits Questionnaire is part of the THINC-Integrated Tool and can be completed in 2-3 minutes. The total score can range between 5 and 25, with higher scores indicating worse outcome (worse cognitive function).
Attention function will be measured in mean latency for correct responses in milliseconds. | Cognitive function, such as attention function will be measured in the first and last week of up to 8-week inpatient treatment.
  Mean latency for correct responses will be tested with the Spotter test, which is part of the THINC-Integrated tool. The Spotter test is inspired by the Choice Reaction Time Test to measure attention function. Higher values indicate worse outcome (worse attention function).
Working memory will be displayed in number of correct responses to the Symbol Check test. | Cognitive function, such as working memory will be measured in the first and last week of up to 8-week inpatient treatment.
  The Symbol Check test is part of the THINC-Integrated Tool and inspired by the One-back test to measure working memory, with higher number of correct responses indicating greater outcome (higher working memory).
Ability to concentrate will be tested with the total number of correct responses to the Codebreaker test. | Cognitive function, such as ability to concentrate will be measured in the first and last week of up to 8-week inpatient treatment.
  The Codebreaker test is part of the THINC-Integrated Tool and inspired by the Digit Symbol Substitution Test to identify the ability to concentrate, with higher number of correct responses indicating greater outcome (better ability to concentrate).
Executive function will be shown in time taken to complete the Trails test in seconds. | Cognitive function, such as executive function will be measured in the first and last week of up to 8-week inpatient treatment.
  The Trails test is part of the THINC-Integrated Tool and inspired by the Trail Making Test to test executive function, with higher values indicating worse outcome (reduced executive function).
Self-reported physical activity, objective measured physical activity and sleep displayed in average minutes per day. | Self-reported physical activity will be screened ones during first week of inpatient treatment. Objective measured physical activity and sleep daily during up to 8-week inpatient treatment.
  Exercise recommendations are expressed in activity intensity and minutes, e.g. 150 minutes of moderate aerobic activity intensity per week.
Balance performance in seconds, tested with a variation of the One-Leg Standing test. | Balance will be measured in the first and last week of up to 8-week inpatient treatment.
  The sum in seconds of the left and right leg will be used to show balance performance, with higher values indicating greater outcome (better balance performance).
Leg strength in time needed to complete the test in seconds, tested with the 10-time chair-rise test. | Leg strength will be measured in the first and last week of up to 8-week inpatient treatment.
  The reciprocal of time needed to complete the test will be multiplied by 100; consequently, good outcome (strength) will be represented by high scores.
Hand grip strength in kg. | Hand grip strength will be assessed in the first and last week of up to 8-week inpatient treatment.
  Handheld dynamometer (Jamar Smart Hand Dynamometer, Performance Health Supply Inc., Cedarburg, USA) will be used to test hand grip strength with higher values indicating greater outcome (higher hand grip strength).
Cardiovascular health will be depicted as brachial systolic and diastolic blood pressure (in mm Hg). | Cardiovascular health, such as brachial systolic and diastolic blood pressure will be assessed in the first and last week of up to 8-week inpatient treatment.
  Oscillometric cuff-based sphygmomanometer on the right arm (Custo screen 310, custo med GmbH, Ottobrunn, Germany) will be used.
Cardiovascular health will be depicted as central systolic and diastolic blood pressure (in mm Hg). | Cardiovascular health, such as central systolic and diastolic blood pressure will be assessed in the first and last week of up to 8-week inpatient treatment.
  Oscillometric cuff-based sphygmomanometer on the right arm (Custo screen 310, custo med GmbH, Ottobrunn, Germany) will be used.
Cardiovascular health will be depicted with pulse wave velocity in m/s. | Cardiovascular health, such as pulse wave velocity will be assessed in the first and last week of up to 8-week inpatient treatment.
  Oscillometric cuff-based sphygmomanometer on the right arm (Custo screen 310, custo med GmbH, Ottobrunn, Germany) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Arno Schmidt-Trucksäss, Prof., Principal Investigator — University of Basel
Locations (1):
- Clinica Holistica Engiadina, Süs, Kanton Graubünden, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Turner W, Bruhl A, Boker H, Schulze B, Marschall K, La Marca R, Pfaff M, Russmann T, Schmidt-Trucksass A. Heart rate vARiability and physical activity in inpatient treatMent of burnOut and DepressIon (HARMODI): protocol of a cross-sectional study with up to 8-week follow up. BMJ Open. 2024 Jun 25;14(6):e081299. doi: 10.1136/bmjopen-2023-081299. PMID 38925684